CLINICAL TRIAL: NCT02437292
Title: Effect of Ischemic Compression With Stretching on Pain Related Parameters in Patients With Upper Back Pain Associated With Myofascial Trigger Point
Brief Title: Effect of Ischemic Compression With Stretching on Patients With Upper Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Vitsarut Buttagat, Dr. Vitsarut Buttagat, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55218152-6
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ischemic compression with stretching (Experimental): The participants will receive the ischemic compression with stretching onto the trapezius muscle
  Interventions: Other: Ischemic compression with stretching
- Control (No Intervention): Rest on the bed

INTERVENTIONS:
Other: Ischemic compression with stretching
  Arms: Ischemic compression with stretching

SUMMARY:
The purpose of this study is to determine the effect of ischemic compression with stretching on pain related parameters including pain intensity, pressure pain threshold, anxiety, cervical range of motion and patient satisfaction in patients with scapular pain associated with myofascial trigger point.

ELIGIBILITY:
Inclusion Criteria:

* The participants have experienced spontaneous upper back pain for longer than 12 weeks (chronic) and that at least one trigger point will be present in the s trapezius muscles. Trigger points will be diagnosed as the presence of focal tenderness in a taut band and with pain recognition.
* The participants will be able to follow instructions.
* Good communication and cooperation.

Exclusion Criteria:

* Fibromyalgia syndrome
* Cervical radiculopathy or myelopathy)
* Cervical spine surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Pain score on Visual analog scale | 5 weeks
  The intensity of pain will be reported by the participant on a visual analog scale ranging from 0 to 10. Zero indicates no pain anywhere and 10 indicates the most pain ever experienced

SECONDARY OUTCOMES:
Pressure Pain Threshold as a measure by pressure algometry | 5 weeks
Anxiety on State Anxiety Inventory | 5 weeks
Cervical range of motion | 5 weeks
Patient satisfaction level | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: VITSARUT BUTTAGAT, Ph.D., Principal Investigator — Mae Fah Luang University